CLINICAL TRIAL: NCT02305966
Title: Evaluation of Implant Fixation in Reverse Total Shoulder Arthroplasty
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, George Athwal, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7519
Record Dates: First submitted 2014-10-30; First posted 2014-12-03 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Arthritis
Keywords: advanced arthritis; shoulder
MeSH Terms: conditions — Arthritis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (4):
- pressfit humerus & non-lateralized glenoid (Active Comparator): All patients will receive a Delta XTEND reverse shoulder implant (DePuy Synthes, Warsaw, IN). At the time of surgery, 0.8 mm diameter Tantalum marker beads will be injected into the bone surrounding the implant, (n = 6 surrounding the glenoid and n = 6 surrounding the proximal humerus). Half of the patients (n = 20) will be randomized by an opaque envelope intra-operatively to receive a cemented humeral component, and half will be randomized to receive a press-fit (uncemented). Similarly, half of the patients (n = 20) will be randomized by an opaque envelope intra-operatively to receive a lateralized glenoid component, and half will be randomized to receive a non-lateralized glenoid component.Therefore, 4 randomization groups will be created and one of them is -pressfit humerus & non-lateralized glenoid.
  Interventions: Procedure: surgery; Device: 0.8 mm diameter Tantalum marker beads
- pressfit humerus & lateralized glenoid (Active Comparator): All patients will receive a Delta XTEND reverse shoulder implant (DePuy Synthes, Warsaw, IN). At the time of surgery, 0.8 mm diameter Tantalum marker beads will be injected into the bone surrounding the implant, (n = 6 surrounding the glenoid and n = 6 surrounding the proximal humerus). Half of the patients (n = 20) will be randomized by an opaque envelope intra-operatively to receive a cemented humeral component, and half will be randomized to receive a press-fit (uncemented). Similarly, half of the patients (n = 20) will be randomized by an opaque envelope intra-operatively to receive a lateralized glenoid component, and half will be randomized to receive a non-lateralized glenoid component.Therefore, 4 randomization groups will be created and one of them is - pressfit humerus & lateralized glenoid.
  Interventions: Procedure: surgery; Device: 0.8 mm diameter Tantalum marker beads
- cemented humerus & non-lateralized glenoid (Active Comparator): All patients will receive a Delta XTEND reverse shoulder implant (DePuy Synthes, Warsaw, IN). At the time of surgery, 0.8 mm diameter Tantalum marker beads will be injected into the bone surrounding the implant, (n = 6 surrounding the glenoid and n = 6 surrounding the proximal humerus). Half of the patients (n = 20) will be randomized by an opaque envelope intra-operatively to receive a cemented humeral component, and half will be randomized to receive a press-fit (uncemented).Similarly, half of the patients (n = 20) will be randomized by an opaque envelope intra-operatively to receive a lateralized glenoid component, and half will be randomized to receive a non-lateralized glenoid component. Therefore, 4 randomization groups will be created and one of them is cemented humerus & non-lateralized glenoid
  Interventions: Procedure: surgery; Device: 0.8 mm diameter Tantalum marker beads
- cemented humerus & lateralized glenoid. (Active Comparator): All patients will receive a Delta XTEND reverse shoulder implant (DePuy Synthes, Warsaw, IN). At the time of surgery, 0.8 mm diameter Tantalum marker beads will be injected into the bone surrounding the implant, (n = 6 surrounding the glenoid and n = 6 surrounding the proximal humerus). Half of the patients (n = 20) will be randomized by an opaque envelope intra-operatively to receive a cemented humeral component, and half will be randomized to receive a press-fit (uncemented).Similarly, half of the patients (n = 20) will be randomized by an opaque envelope intra-operatively to receive a lateralized glenoid component, and half will be randomized to receive a non-lateralized glenoid component.Therefore, 4 randomization groups will be created and one of them is cemented humerus & lateralized glenoid.
  Interventions: Procedure: surgery; Device: 0.8 mm diameter Tantalum marker beads

INTERVENTIONS:
Procedure: surgery — All patients will receive a Delta XTEND reverse shoulder implant
Device: 0.8 mm diameter Tantalum marker beads — At the time of surgery, 0.8 mm diameter Tantalum marker beads will be injected into the bone surrounding the implant,

SUMMARY:
Reverse total shoulder replacement surgery (RTSA) is performed for individuals with advanced arthritis of the shoulder who also have tears in their rotator cuff muscles. A metal hemisphere is placed in the shoulder blade, and a plastic cup on a stem is placed in the upper arm. This orientation is opposite to the normal anatomy, giving rise to the term "reverse" shoulder replacement. While RTSA has a good clinical track record, no studies have examined how well fixed the implanted components are within patients.

ELIGIBILITY:
Inclusion Criteria:

* will be any patient with cuff tear arthropathy requiring reverse shoulder arthroplasty.

Exclusion Criteria:

* will be any patient with a previous RTSA or TSA (i.e. no revision surgery) or anyone unable to return for RSA imaging (e.g. living >100 km outside of London).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
migration between cemented and press-fit RTSA humeral components detected by Radiostereometric analysis | 24 months

SECONDARY OUTCOMES:
difference in component migration between conventional and lateralized glenoid components detected by Radiostereometric analysis | 24 months